CLINICAL TRIAL: NCT03892395
Title: A Randomised Controlled Trial to Investigate the Effect of Combined B-vitamin Supplementation for 2-years on Bone Mineral Density in Older Irish Adults With Sub-optimal B-vitamin Status
Brief Title: An Intervention Study to Investigate the Effect of B-vitamin Supplementation for 2-years on Bone Health
Acronym: Opti-Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: University of Ulster (Other)
Responsible Party: Principal Investigator, Lorraine Brennan, Principle Investigator, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UCD_456_2019
Record Dates: First submitted 2019-03-22; First posted 2019-03-27 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Bone Health
Keywords: Healthy ageing; B-vitamins; Bone health
MeSH Terms: interventions — Control Groups; Vitamin D

STUDY DESIGN:
Intervention Model Description: Supplementation for 2 years with one of the following treatments in capsule form:
  1. Active: B vitamins + vitamin D, a daily capsule containing 200 µg/day folic acid, 10 µg/day vitamin B12, 10 mg/day vitamin B6 and 5 mg/day riboflavin, and 10 µg/day vitamin D combined.
  2. Control/Placebo: Vitamin D, a daily capsule containing 10 µg/day vitamin D
Who Masked: Participant, Investigator
Masking Description: 2 year randomised, placebo controlled, double blinded intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Supplementation for 2 years with one of the following treatments in capsule form:
  Treatment group will receive: B vitamins + vitamin D, a daily capsule containing 200 µg/day folic acid, 10 µg/day vitamin B12, 10 mg/day vitamin B6 and 5 mg/day riboflavin, and 10 µg/day vitamin D combined
  Interventions: Dietary Supplement: B-vitamin supplementation on bone health
- Control group (Placebo Comparator): Supplementation for 2 years with one of the following treatments in capsule form:
  Control group will receive: Vitamin D, a daily capsule containing 10 µg/day vitamin D
  Interventions: Dietary Supplement: Control group; Vitamin D, a daily capsule containing 10 µg/day vitamin D

INTERVENTIONS:
Dietary Supplement: B-vitamin supplementation on bone health — An intervention study to investigate the effect of B-vitamin supplementation for 2-years on bone health
  Arms: Treatment group
Dietary Supplement: Control group; Vitamin D, a daily capsule containing 10 µg/day vitamin D — Vitamin D, a daily capsule containing 10 µg/day vitamin D
  Arms: Control group

SUMMARY:
An intervention study to investigate the effect of B-vitamin supplementation for 2-years on bone health. This is a dual centre (UCD and University of Ulster) 2-year randomised, placebo controlled, double blind intervention.

DETAILED DESCRIPTION:
Osteoporosis is a major public health issue, especially among older adults. The condition is widespread, with an estimated 1 in 2 women and 1 in 5 men over the age of 50 years expected to have an osteoporotic fracture. The associated health care costs are considerable and growing as the population of older adults increases. Furthermore, osteoporotic fractures are associated with loss of independence and risk of further fractures and health problems for the individual. Given these negative impacts, new approaches to help maintain better bone health in older age are urgently needed.

Vitamin D and calcium have well established protective roles, however, other evidence links certain B vitamins with bone health. This study will investigate the effect of B-vitamin supplementation over a two year period at two centres (UCD and University of Ulster)

ELIGIBILITY:
Inclusion Criteria:

* 50 years and over
* Generally healthy, free living in the community
* Males and females (post menopausal and not taking HRT)

Exclusion Criteria:

* Currently taking a supplement containing B vitamins
* Currently consuming >4 portions of foods fortified with B vitamins per week
* Currently taking drugs known to interfere with folate/ B-vitamin metabolism
* Have a condition of the gastrointestinal system (such as coeliac disease/ chron's disease, ulcerative colitis) or liver disease (hepatitis and NAFLD)
* Be unable to consent to participate
* Be currently involved in another research study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Effect of low dose B vitamins on bone mineral density | 2 years
  A 2 year Randomized Control Trial (RCT) to investigate the effect of low dose B vitamins on bone mineral density (as measured by dual energy X-ray absorptiometry- DXA) in older Irish adults with sub-optimal B-vitamin status at baseline. A DXA bone scan will be performed pre and post the 2-year intervention to evaluate beneficial effects to bone mineral density

SECONDARY OUTCOMES:
Metabolomics | 2 years
  Metabolomics analysis of blood samples collected pre and post the trial to explore the mechanistic effects of B- vitamins on bone and other outcomes
Neurocognitive function I | 2 years
  To determine the neurocognitive function using the Mini Mental State Exam 'MMSE' test (pre- and post-intervention)
Neurocognitive function II | 2 years
  To determine the neurocognitive function using the Repeatable Battery for the Assessment of Neuropsychological Status 'RBANS' test (pre- and post-intervention)
Neurocognitive function III | 2 years
  To determine the neurocognitive function using the Frontal Assessment Battery 'FAB' test (pre- and post-intervention)
Gut microbiome | 2 years
  To collect faecal samples pre and post intervention to explore potential interactions with the gut microbiome
Blood pressure | 2 years
  To measure blood pressure throughout the study and compare baseline to post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Brennan, PhD, Principal Investigator — University College Dublin
Locations (1):
- University College Dublin, Dublin, Dublin 4, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clements M, Heffernan M, Ward M, Hoey L, Doherty LC, Hack Mendes R, Clarke MM, Hughes CF, Love I, Murphy S, McDermott E, Grehan J, McCann A, McAnena LB, Strain JJ, Brennan L, McNulty H. A 2-Year Randomized Controlled Trial With Low-Dose B-Vitamin Supplementation Shows Benefits on Bone Mineral Density in Adults With Lower B12 Status. J Bone Miner Res. 2022 Dec;37(12):2443-2455. doi: 10.1002/jbmr.4709. Epub 2022 Oct 14. PMID 36128889